CLINICAL TRIAL: NCT00376584
Title: A Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Study to Evaluate the Efficacy of MK0524 to Improve Tolerability of Extended Release Niacin
Brief Title: Effect of an Investigational Compound on Tolerability of Extended Release Niacin (0524A-023)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-023; MK0524A-023; 2006_504
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Hypercholesteremia; Hyperlipidemia
Keywords: Primary Hypercholesteremia; Mixed Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo → MK-0524A 2g (Placebo Comparator): Following an 8-week active run-in (MK-0524A 1g (4 Weeks) then MK-0524A 2g (4 weeks) participants will be administered MK-0524A Placebo for 5 days (drug holiday) followed by MK-0524A 2 g for the remainder of the study (7 days).
  Interventions: Drug: MK-0524A; Drug: Placebo
- Placebo → Extended Release (ER)-Niacin 2g (Active Comparator): Following an 8-week active run-in (MK-0524A 1g (4 Weeks) then MK-0524A 2g (4 weeks) participants will be administered MK-0524A Placebo for 5 days (drug holiday) followed by ER-Niacin 2g for the remainder of the study (7 days)
  Interventions: Drug: ER Niacin; Drug: Placebo
- MK-0524A 2g (Experimental): Following an 8-week active run-in (MK-0524A 1g (4 Weeks) then MK-0524A 2g (4 weeks) participants will be administered MK-0524A 2g for the remainder of the study (approximately 2 weeks).
  Interventions: Drug: MK-0524A

INTERVENTIONS:
Drug: MK-0524A
  Arms: MK-0524A 2g; Placebo → MK-0524A 2g
Drug: ER Niacin
  Arms: Placebo → Extended Release (ER)-Niacin 2g
Drug: Placebo
  Arms: Placebo → Extended Release (ER)-Niacin 2g; Placebo → MK-0524A 2g

SUMMARY:
This is a 12-week clinical trial in lipid clinic patients for whom niacin therapy is appropriate to evaluate the efficacy of MK0524 to improve the tolerability of extended-release niacin. There will be 6 scheduled clinic visits and 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patient is appropriate candidate for niacin therapy
* Patients with evidence of ischemic cardiovascular disease must be on a statin and have LDL-C <130 mg/dL at V1
* Patients with diabetes mellitus and no evidence of ischemic cardiovascular disease must have LDL-C <130 mg/dL at V1
* Non-diabetic patients with 2 or more risk factors for coronary heart disease and no ischemic cardiovascular disease must have LDL-C <160 mg/dL at V1
* Patient has TG <500 mg/dL (5.65 mmol/L) at V1
* A patients historic serum or plasma lipid values measured within 6 months from Visit 1 may be used to meet lipid inclusion criteria
* ALL OTHER PATIENTS DO NOT REQUIRE SPECIFIC LIPID ENTRY CRITERIA

Exclusion Criteria:

* Patients with unstable doses of medications
* Pregnant or lactating women, or women intending to become pregnant are excluded
* Patients with diabetes mellitus that is poorly controlled, unstable or newly diagnosed
* Patients with: chronic heart failure, uncontrolled/unstable cardiac arrhythmias, unstable hypertension, active or chronic hepatobiliary disorder or hepatic disease, HIV positive, gout (within 1 year)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2006-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Global Flushing Severity Score (GFSS) during 7 days of treatment | during 7 days of treatment

SECONDARY OUTCOMES:
Percentage of Participants Who Experience at Least 1 Adverse Event | up to 10 weeks
Percentage of Participants Who Were Discontinued from the Study Due to an Adverse Event | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html